CLINICAL TRIAL: NCT04389567
Title: Famotidine Use in Non-hospitalized Patients With COVID-19: A Case Series
Brief Title: Famotidine Outpatient COVID-19 Treatment Study
Status: Completed | Type: Observational
Sponsor: Northwell Health (Other)
Collaborators: Cold Spring Harbor Laboratory (Other)
Responsible Party: Sponsor
Other Study IDs: 1605914-1
Record Dates: First submitted 2020-05-13; First posted 2020-05-15 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: COVID-19
Keywords: Famotidine
MeSH Terms: conditions — COVID-19 | interventions — Famotidine

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with COVID-19 taking Famotidine: Use of any dose of oral Famotidine during period of COVID-19
  Interventions: Drug: Famotidine

INTERVENTIONS:
Drug: Famotidine — Use of oral Famotidine.

SUMMARY:
A retrospective case series of patients who self-medicated with Famotidine during coronavirus disease 2019 (COVID-19). The study will collect de-identified patient reported outcome measures of patients with confirmed COVID-19 who self-medicated with Famotidine at any dose during the period of illness. Data will be collected by questionnaire and telephone interview.

Inclusion criteria:

Age>18; Ability to give written informed consent for study participation; Confirmed diagnosis of COVID-19; Use of Famotidine at any dose during period of COVID-19 illness

DETAILED DESCRIPTION:
Famotidine is a histamine-2 receptor antagonist, widely available over-the-counter, and is safely used for suppression of gastric acid production over a wide range of doses from 20mg once daily to 160mg four times daily. In computer-based simulations, Famotidine has been identified as a potential inhibitor of the 3-chymotrypsin-like protease (3CLpro). In a propensity score matched retrospective cohort study a significantly reduced risk for death or intubation (adjusted hazard ratio 0.43, 95% confidence interval 0.21-0.88) was identified for patients with COVID-19 who were taking Famotidine before or at the point of hospital admission. Some individuals have self-medicated with Famotidine while being outpatients with COVID-19. This study is aimed at collecting patient reported outcome measures from such individuals.

ELIGIBILITY:
Inclusion Criteria:

Age >18 years; Ability to give written informed consent; Confirmed COVID-19 diagnosis; Famotidine use during COVID-19 illness

Exclusion Criteria:

none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study allows participants from all demographics.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2020-05-12 (Actual); Primary Completion 2020-05-25 (Actual); Study Completion 2020-05-25 (Actual)

PRIMARY OUTCOMES:
Symptomatic improvement | 2 weeks
  Symptoms assessed by severity scores on an ordinal scale; 1=not affected to 4= severely affected

SECONDARY OUTCOMES:
Peripheral blood oxygen saturation | 2 weeks
  Oxygen saturation determined by pulse oximetry

CONTACTS AND LOCATIONS:
Overall Officials: David A Tuveson, MD PhD, Principal Investigator — Cold Spring Harbor Laboratory
Locations (1):
- Cold Spring Harbor Laboratory, Cold Spring Harbor, New York, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared with other researchers. De-identified data will be reported in a case series publication. All participants have consented to having de-identified data included in a case series report.

REFERENCES:
- [Background] Wu C, Liu Y, Yang Y, Zhang P, Zhong W, Wang Y, Wang Q, Xu Y, Li M, Li X, Zheng M, Chen L, Li H. Analysis of therapeutic targets for SARS-CoV-2 and discovery of potential drugs by computational methods. Acta Pharm Sin B. 2020 May;10(5):766-788. doi: 10.1016/j.apsb.2020.02.008. Epub 2020 Feb 27. PMID 32292689
- [Background] Freedberg DE, Conigliaro J, Wang TC, Tracey KJ, Callahan MV, Abrams JA; Famotidine Research Group. Famotidine Use Is Associated With Improved Clinical Outcomes in Hospitalized COVID-19 Patients: A Propensity Score Matched Retrospective Cohort Study. Gastroenterology. 2020 Sep;159(3):1129-1131.e3. doi: 10.1053/j.gastro.2020.05.053. Epub 2020 May 22. No abstract available. PMID 32446698